CLINICAL TRIAL: NCT00204373
Title: Long-Term Study of the Efficacy and Safety of Lansoprazole in the Treatment of Zollinger-Ellison and Other Acid Hypersecretors
Brief Title: Treatment of Zollinger-Ellison Syndrome With Prevacid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Mel Wilcox, MD (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Charles Mel Wilcox, MD, Prinicle Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F030107005
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Zollinger-Ellison Syndrome; Multiple Endocrine Neoplasia
MeSH Terms: conditions — Zollinger-Ellison Syndrome; Multiple Endocrine Neoplasia | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single group (Experimental): This is an open label, non-randomized, uncontrolled, single group study designed to treat patients with Zollinger-Ellison Syndrome and other hypersecretory conditions by controlling gastric acid production; to heal and prevent relapses of peptic ulcers and symptoms; to monitor the safety and efficacy of this treatment.
  Interventions: Drug: Lansoprazole (Prevacid)

INTERVENTIONS:
Drug: Lansoprazole (Prevacid) — Lansoprazole 30mg capsules. dose is individualized to each subject based on gastric acid production. The range is 30 mg to 450 mg daily.
  Other Names: Lansoprazole is marketed as Prevacid.

SUMMARY:
The purpose of this study is to study the safety and efficacy of high dose Prevacid in the long-term treatment of patients who secrete abnormally large amounts of gastric acid.

DETAILED DESCRIPTION:
The aim of this protocol is to study the medical management of acid hypersecretory states including Zollinger-Ellison using Prevacid. The immediate objective is to heal peptic ulcers and eliminate symptoms and in the long term to prevent relapse of symptoms, lesions and complications. Other objectives include observation of the efficacy in controlling gastric acid production and of the safety of high dose, long-term use of Prevacid.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Zollinger-Ellison syndrome

Exclusion Criteria:

* Pregnant or lactating females

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Mel Wilcox, M.D., Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Result] Hirschowitz BI, Simmons J, Mohnen J. Clinical outcome using lansoprazole in acid hypersecretors with and without Zollinger-Ellison syndrome: a 13-year prospective study. Clin Gastroenterol Hepatol. 2005 Jan;3(1):39-48. doi: 10.1016/s1542-3565(04)00606-8. PMID 15645403
- [Result] Wilcox CM, Seay T, Arcury JT, Mohnen J, Hirschowitz BI. Zollinger-Ellison syndrome: presentation, response to therapy, and outcome. Dig Liver Dis. 2011 Jun;43(6):439-43. doi: 10.1016/j.dld.2010.11.007. Epub 2010 Dec 30. PMID 21193359
- [Derived] Wilcox CM, Seay T, Arcury J, Hirschowitz BI. Presentation, response to lansoprazole therapy, and outcome of Zollinger-Ellison syndrome-like gastric acid hypersecretors. Scand J Gastroenterol. 2011 Mar;46(3):277-80. doi: 10.3109/00365521.2010.536255. Epub 2010 Nov 15. PMID 21073392
- [Derived] Hirschowitz BI, Fineberg N, Wilcox CM, Mohnen J, Worthington J. Costs and risks in the management of patients with gastric acid hypersecretion. J Clin Gastroenterol. 2010 Jan;44(1):28-33. doi: 10.1097/MCG.0b013e3181a59aa5. PMID 19581810
- [Derived] Wilcox CM, Martin T, Phadnis M, Mohnen J, Worthington J, Hirschowitz BI. Absence of gastrointestinal infections in a cohort of patients with Zollinger-Ellison syndrome and other acid hypersecretors receiving long-term acid suppression with lansoprazole. BMC Gastroenterol. 2008 May 28;8:18. doi: 10.1186/1471-230X-8-18. PMID 18507843
- [Derived] Hirschowitz BI, Worthington J, Mohnen J, Haber M. Chromogranin A in patients with acid hypersecretion and/or hypergastrinaemia. Aliment Pharmacol Ther. 2007 Sep 15;26(6):869-78. doi: 10.1111/j.1365-2036.2007.03439.x. PMID 17767471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the GI/Hepatology clinic located at The Kirklin Clinic. Patients were referred here from their primary care physician or chose this clinic through self-referral for care for a GI issue. Patients were recruited between early 2003 and early 2010.
Pre-assignment Details: The first phase of this study involved a short-term dose determination phase followed by a long-term treatment phase.
Period: Overall Study
Arm/Group | Single Group
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Group
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Long-term Medical(Non-surgical)Control of Gastric Acid Production Assessed From Time of Study Enrollment, up to 240 Months Post Enrollment.
Description: number of participants with control of gastric acid production
Time Frame: up to 240 months from study enrollment
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 72
participants | 72

2. Secondary Outcome: The Median Survival From the Time of Diagnosis.
Description: The median survival from the time of diagnosis
Time Frame: survival or up to 240 months
Measure: Median (Standard Deviation); unit: years
Arm/Group | Single Group
Number analyzed (Participants) | 72
years | 6.6 (1.8)

ADVERSE EVENTS:
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 28/72
Other Adverse Events (participants affected / at risk) | 21/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group (N=72)
Mucosal relapse (Gastrointestinal disorders) | 12 (12) — Mucosal relapse was documented in 12 pts (16.7%). The type or relapse included a peptic ulcer in 4.2% (0 gastric, 3 duodenal), reflux oesophagitis in 8 (11.1%) and small bowel perforation in 2 (2.8%).
Death (Cardiac disorders) | 9 (9) — The most common cause of death was cardiovascular disease or stroke (9 pts).
Cancer (Gastrointestinal disorders) | 5 (5) — 5 patients developed cancer including pancreatic, gallbladder and lung cancers.
Death (metastatic gastrinoma) (Gastrointestinal disorders) | 2 (2) — Two patients died due to progressive metastatic gastrinoma.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group (N=72)
Nausea and vomiting (Gastrointestinal disorders) | 13 (13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Leg Pain (Musculoskeletal and connective tissue disorders) | 4 (4) — 4 patients experienced leg pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No